CLINICAL TRIAL: NCT05286216
Title: The Effect of Education on Oral Antiviral Use on Medication Compliance and Quality of Life in Patients With Hepatitis-B Diagnosis
Brief Title: The Effect of Education on Drug Compliance and Quality of Life in Hepatitis B Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sengul KORKMAZ BINAY, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sengul Korkmaz Binay Tez
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B, Chronic; Adherence, Medication; Quality of Life
Keywords: chronic hepatitis B; adherence, medication; quality of life
MeSH Terms: conditions — Hepatitis B, Chronic; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient diagnosis form with CHB and related scales (Patient Diagnosis Form with Chronic Hepatitis B, Medication Adherence Report Scale-5), Medication Adherence Report Scale (MedTake Test), Chronic Liver Disease Quality of Life Scale 2.0" (Liver Disease Symptom Index 2.0 (LDSI 2.0), Health-Related Quality of Life Scale SF-12" (12 Item Short Form Health Survey) (Short Form 12 - SF 12), Patient Learning Needs Scale will be applied before the intervention. The training will be in two modules and two different sessions. The effectiveness of the training will be evaluated by re-applying the scales 12 weeks and 24 weeks after the training.
  Interventions: Behavioral: effectiveness of education
- Control group (No Intervention): Patient diagnosis form with CHB and related scales (Patient Diagnosis Form with Chronic Hepatitis B, Medication Adherence Report Scale-5), Medication Adherence Report Scale (MedTake Test), Chronic Liver Disease Quality of Life Scale 2.0" (Liver Disease Symptom Index 2.0 (LDSI 2.0), Health-Related Quality of Life Scale SF-12" (12 Item Short Form Health Survey) (Short Form 12 - SF 12), Patient Learning Needs Scale in the first evaluation, 12 weeks and 24 weeks later, the scales were re-applied and the education was improved. effectiveness will be evaluated.

INTERVENTIONS:
Behavioral: effectiveness of education — The education program will be prepared using power point presentations within the relevant scientific literature. The education program is planned to be given to each group as 1 session on 2 different days, between 09:30 and 13:00. Day 1 module 1; Module 2 will be shared on the 2nd day and all patients in the experimental group will participate in the education program. During and after the education, individuals will be provided with the opportunity to ask questions. In addition, after the education, the researcher's phone will be given and counseling will be provided by phone. The duration and subject of the telephone conversations will be recorded by the researcher.
  In order to evaluate the training, all patients will be invited to the hospital on the day of the control at the end of 12 and 24 weeks, and evaluations will be made again with data collection tools.
  Arms: Experimental group

SUMMARY:
The aim of this study is to determine the effect of the education given to patients with CHB who use oral antiviral drugs on oral antiviral drug use on drug compliance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with CHB for at least 6 months,

  * To be over 18 years old,
  * Using oral antiviral treatment for at least three months,
  * To be a literate person,
  * No malignancy other than hepatocellular carcinoma,
  * Not having vision and hearing problems,
  * Not having cognitive or psychiatric problems,
  * Patients/patient relatives who can use smartphones (In order to invite the patients to the 3rd and 6th month controls and to inform and remind the experimental group about the training time, they / their relatives should have and can use a mobile phone)
  * Volunteer to participate in the study.

Exclusion Criteria:

* •Continuing to use alcohol after the first evaluation,

  * Not willing to participate in the study,
  * Patients with a psychiatric diagnosis,
  * Patients who do not meet the sample inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Report Scale-5 | 24 weeks
  Medication Adherence Report Scale-5: Scores from the 5-point Likert-type scale vary between 5 and 25. An increase in the obtained scores indicates compatibility, and a decrease in scores indicates inconsistency.
MedTake Test | 24 weeks
  MedTake Test: It is used to evaluate the use of prescribed oral drugs and to numerically show patients' compliance with drug treatments. With the scale, the daily dose, time and frequency of taking the drug, its effect and reason for taking it, and its relationship with food (hungry-full) are evaluated for each drug. For these 4 parameters, patients score out of 25. In total, the level of knowledge for each drug is scored out of 100. Compliance score for all treatments is calculated with all scores of the patients. Compliance score of the participants in the study is calculated with the total compliance score obtained by each participant.
Liver Disease Symptom Index 2.0 | 24 weeks
  Liver Disease Symptom Index 2.0: The scale is divided into two parts and includes 24 questions in total. The first part consists of a total of 18 questions, 9 main and 9 sub-questions, questioning the effects of the disease in the last 1 week, and the second part consists of 6 main questions questioning the effects of the disease from the time the patient learned about the disease to the present. The answer to each question in the scale receives a score between a minimum of '1' and a maximum of '5'. '1' is the lowest score; '5' represents the highest score. Higher scores from the scale indicate worse quality of life.
Composite 12 İtem Short Form Health Survey | 24 weeks
  Composite 12 İtem Short Form Health Survey: It has a physical and mental component. Both the Physical Component Scale-12 and the Mental Component Scale-12 scores range from 0 to 100, with a higher score indicating better health.

IPD SHARING:
Plan to Share IPD: No